CLINICAL TRIAL: NCT00503113
Title: A Randomized, Open Label Study Evaluating the Effect on Renal Function of Intravenous Bonviva Given by Injection or Infusion, Compared With Oral Alendronate, in Postmenopausal Women With Osteoporosis at High Risk for Renal Disease.
Brief Title: A Study of Bonviva (Ibandronate) and Alendronate on Renal Function in Postmenopausal Women With Osteoporosis at High Risk for Renal Disease.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Disclosures Group, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BA20341
Record Dates: First submitted 2007-07-17; First posted 2007-07-18 (Estimated); Results first posted 2011-06-17 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-05

CONDITIONS: Post-Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid; Alendronate

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Experimental)
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 3 (Active Comparator)
  Interventions: Drug: Alendronate

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 3mg intravenous (iv) injection every 3 months
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 3mg intravenous (iv) infusion every 3 months
  Arms: 2
Drug: Alendronate — 70mg per oral (po) weekly
  Arms: 3

SUMMARY:
This 3 arm study will evaluate renal safety after administration of an intravenous (iv) injection or infusion of Bonviva, compared to oral alendronate, in patients with postmenopausal osteoporosis, at increased risk of renal disease. Patients will be randomized to receive Bonviva 3mg intravenous (iv) by a) injection or b) infusion once every 3 months, or alendronate 70mg per oral (po) weekly. The anticipated time on study treatment is 3-12 months, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=60 years of age;
* >=5 years postmenopausal;
* confirmed osteoporosis, at increased risk for renal disease.

Exclusion Criteria:

* inability to stand or sit upright for 30 minutes;
* hypersensitivity to bisphosphonates;
* malignant disease (other than successfully resected basal cell cancer) within previous 10 years, or breast cancer diagnosed within previous 20 years;
* previous administration of an i.v. bisphosphonate;
* oral bisphosphonate treatment other than study medication within 30 days prior to the baseline dosing visit and during the study;
* history of major upper gastrointestinal disease.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801 (Actual)
Dates: Start 2007-07; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (38):
- United States (15):
  - Birmingham, Alabama
  - Riverside, California
  - Lakewood, Colorado
  - West Palm Beach, Florida
  - Gainesville, Georgia
  - Topeka, Kansas
  - Bethesda, Maryland
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - Morehead City, North Carolina
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Duncansville, Pennsylvania
  - Norfolk, Virginia
- Argentina (3):
  - Buenos Aires
  - Córdoba
  - Santa Fe
- Brazil (7):
  - Brasília
  - Curitiba
  - Goiânia
  - Porto Alegre
  - Rio de Janeiro
  - São Paulo
  - Vitória
- Mexico (5):
  - Guadalajara
  - Mexico City
  - Monterrey
  - Obregón
  - San Jerónimo
- South Africa (5):
  - Durban
  - Johannesburg
  - Parow
  - Port Elizabeth
  - Somerset West
- Switzerland (3):
  - Basel
  - Bern
  - Zurich

REFERENCES:
- [Derived] Hara T, Hijikata Y, Matsubara Y, Watanabe N. Pharmacological interventions versus placebo, no treatment or usual care for osteoporosis in people with chronic kidney disease stages 3-5D. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013424. doi: 10.1002/14651858.CD013424.pub2. PMID 34231877

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 801 participants randomized. Of the randomized patients, 263 who received at least one dose of ibandronate as an injection, 263 who received at least one dose of ibandronate as an infusion and 267 patients who received at least one dose of alendronate had at least one post-baseline assessment and were included in the safety analysis.
Groups:
- Ibandronate 3 mg Injection: Ibandronate was administered as an intravenous (iv) injection (15 to 30 seconds) of 3 mg every 3 months.
- Ibandronate 3 mg Infusion: Ibandronate was administered as an intravenous (iv) infusion (15 min) of 3 mg every 3 months.
- Alendronate 70 mg Oral: Alendronate was administered as an oral tablet of 70 mg every week (Fosamax 70 mg).
Period: Overall Study
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Started | 268 | 264 | 269
Intent to Treat Population (ITT) | 262 | 261 | 268
Per Protocol Population (PP) | 246 | 243 | 241
Safety Population | 263 | 263 | 267
Completed | 235 | 236 | 241
Not Completed | 33 | 28 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral | Total
Number analyzed (Participants) | 263 | 263 | 267 | 793
Age Continuous [Mean (Standard Deviation); unit: years] | 71.7 (6.77) | 71.5 (5.89) | 71.7 (6.3) | 71.6 (6.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 263 | 267 | 793
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Actual Glomerular Filtration Rate (GFR) (Using Abbreviated Modification of Diet in Renal Disease [MDRD] Formula)
Description: The primary parameter of the study was the change (mL/min) from baseline in actual GFR (abbreviated MDRD formula using the patients' actual body surface area) after 9 months (or 40 weeks) of treatment.
Time Frame: Baseline and 9 months
Population: Per Protocol (PP) Population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mL/min
  Baseline | 72.5 (18.25) | 71.5 (18.07) | 70.5 (16.67)
  Change from baseline at 9 months (n=233,232,225) | -1.3 (7.14) | -0.5 (7.86) | -1.6 (5.89)

2. Secondary Outcome: Absolute Change From Baseline in Actual GFR (Using Cockcroft-Gault [CG] Formula)
Description: Change (mL/min) from baseline in actual GFR (using Cockcroft-Gault [CG] formula) after 9 months (or 40 weeks) of treatment.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mL/min
  Baseline | 65.0 (19.37) | 62.9 (18.22) | 62.0 (16.67)
  Change from Baseline at 9 months (N=233,232,225) | -1.6 (5.89) | -1.0 (6.44) | -1.9 (4.84)

3. Secondary Outcome: Relative Change From Baseline in Actual GFR (Using Abbreviated MDRD Formula)
Description: Change (mL/min) from baseline in actual GFR (abbreviated MDRD formula using the patient's actual body surface area) after 9 months (or 40 weeks) of treatment.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mL/min
  Baseline | 72.5 (18.25) | 71.5 (18.07) | 70.5 (16.67)
  Relative Change at 9 month (n= 233, 232, 225) | -1.4 (10.01) | -0.2 (10.73) | -2.1 (8.64)

4. Secondary Outcome: Relative Change From Baseline in Actual GFR (Using CG Formula)
Description: Change (mL/min) from baseline in actual GFR (CG formula using the patient's actual body surface area) after 9 months (or 40 weeks) of treatment.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mL/min
  Baseline | 65.0 (19.37) | 62.9 (18.22) | 62.0 (16.76)
  Relative Change at 9 month (n=233,232,225) | -2.3 (9.22) | -1.3 (9.55) | -2.8 (7.97)

5. Secondary Outcome: Absolute Change From Baseline in Mean Serum Creatinine.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mg/dL
  Baseline | 0.8 (0.17) | 0.8 (0.16) | 0.8 (0.16)
  Change from Baseline at 9 months (n=233,232,225) | 0.0 (0.08) | 0.0 (0.08) | 0.0 (0.07)

6. Secondary Outcome: Relative Change From Baseline in Mean Serum Creatinine.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mg/dL
  Baseline | 0.8 (0.17) | 0.8 (0.16) | 0.8 (0.16)
  Relative Change at 9 months (n=233,232,225) | 1.7 (8.87) | 0.8 (8.87) | 2.2 (8.06)

7. Secondary Outcome: Absolute Change From Baseline in Urine Albumin-to-Creatinine Ratio.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mg/g
  Baseline | 16.0 (17.30) | 14.1 (15.22) | 16.1 (19.11)
  Change from Baseline at 9 months (n=233,232,225) | -0.8 (18.54) | 0.5 (14.70) | 1.4 (22.99)

8. Secondary Outcome: Relative Change From Baseline in Urine Albumin-to-Creatinine Ratio.
Description: The relative change from baseline in this case is positively skewed (while the absolute change is not) and the means tends to more positive values.
Time Frame: Baseline and 9 months
Population: PP Population
Measure: Mean (Standard Deviation); unit: mg/g
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Number analyzed (Participants) | 246 | 243 | 241
mg/g
  Baseline | 16.0 (17.30) | 14.1 (15.22) | 16.1 (19.11)
  Relative Change at 9 month (n=233,232,225) | 21.6 (120.98) | 15.6 (62.32) | 28.3 (116.71)

ADVERSE EVENTS:
Time Frame: AEs are considered to have occurred 'On treatment', defined as first dose and up 106 days after last dose if patient's actual treatment is ibandronate, or up to 22 days after last dose if patient's actual treatment is the alendronate.
Arm/Group | Ibandronate 3 mg Injection | Ibandronate 3 mg Infusion | Alendronate 70 mg Oral
Serious Adverse Events (participants affected / at risk) | 19/263 | 15/263 | 13/267
Other Adverse Events (participants affected / at risk) | 196/263 | 190/263 | 191/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 3 mg Injection (N=263) | Ibandronate 3 mg Infusion (N=263) | Alendronate 70 mg Oral (N=267)
Femur Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 4
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Multiple Drug Overdose Accidental (Injury, poisoning and procedural complications) | 0 | 0 | 1
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac Failure Congestive (Cardiac disorders) | 2 | 0 | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 1 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0
Conduction Disorder (Cardiac disorders) | 0 | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 1
Abdominal Abscess (Infections and infestations) | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 1 | 0 | 0
Peptic Ulcer Perforation (Gastrointestinal disorders) | 0 | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Breast Cancer Stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0
Ischemic Stroke (Nervous system disorders) | 1 | 0 | 0
Ruptured Cerebral Aneurysm (Nervous system disorders) | 0 | 0 | 1
Senile Dementia (Nervous system disorders) | 0 | 1 | 0
Subarachnoid Haemorrhage (Nervous system disorders) | 1 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 1
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1 | 0
Temporal Arteritis (Vascular disorders) | 0 | 1 | 0
Autoimmune Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0
Electrolyte Imbalance (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Breast Mass (Reproductive system and breast disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 3 mg Injection (N=263) | Ibandronate 3 mg Infusion (N=263) | Alendronate 70 mg Oral (N=267)
Influenza (Infections and infestations) | 37 | 32 | 30
Back Pain (Musculoskeletal and connective tissue disorders) | 26 | 29 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 28 | 27
Hypertension (Vascular disorders) | 23 | 28 | 16
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 22 | 23 | 21
Myalgia (Musculoskeletal and connective tissue disorders) | 22 | 14 | 6
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 19 | 15 | 7
Dizziness (Nervous system disorders) | 19 | 12 | 9
Diarrhoea (Gastrointestinal disorders) | 7 | 11 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 5 | 17
Headache (Nervous system disorders) | 14 | 15 | 6
Dyspepsia (Respiratory, thoracic and mediastinal disorders) | 5 | 11 | 17
Nasopharyngitis (Infections and infestations) | 12 | 12 | 8
Bronchitis (Infections and infestations) | 10 | 11 | 10
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 9 | 13
Influenza Like Illness (General disorders) | 15 | 14 | 1
Nausea (Gastrointestinal disorders) | 10 | 10 | 10
Oedema Peripheral (General disorders) | 12 | 6 | 12
Urinary Tract Infection (Infections and infestations) | 9 | 10 | 11
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 6 | 7 | 13
Anxiety (Psychiatric disorders) | 5 | 10 | 10
Depression (Psychiatric disorders) | 11 | 8 | 5
Fall (Injury, poisoning and procedural complications) | 13 | 8 | 3
Gastroenteritis (Infections and infestations) | 3 | 11 | 9
Anaemia (Blood and lymphatic system disorders) | 8 | 9 | 5
Constipation (Gastrointestinal disorders) | 8 | 9 | 5
Dyslipidemia (Metabolism and nutrition disorders) | 2 | 8 | 10
Gastritis (Gastrointestinal disorders) | 5 | 8 | 7
Upper Respiratory Tract Infection (Infections and infestations) | 5 | 7 | 8
Vomiting (Gastrointestinal disorders) | 8 | 7 | 4
Sciatica (Nervous system disorders) | 6 | 7 | 5
Abdominal Pain (Gastrointestinal disorders) | 6 | 7 | 4
Pain (General disorders) | 6 | 9 | 2
Bone Pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 2
Glomerular Filtration Rate Decreased (Investigations) | 2 | 3 | 11
Labyrinthitis (Infections and infestations) | 7 | 3 | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 6 | 5 | 5
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 6 | 0 | 8
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 4 | 7
Sinusitis (Infections and infestations) | 4 | 4 | 6
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 2
Haemorrhoids (Gastrointestinal disorders) | 7 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No